CLINICAL TRIAL: NCT05706363
Title: Comparison of Two Graft Choices in Mediale Patellofemoral Ligament Reconstruction (MPFL) - A Randomized Controlled Trial.
Brief Title: Comparison of Two Graft Choices in Mediale Patellofemoral Ligament Reconstruction (MPFL)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Martin Lind, Professor, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Danish EC: 1-10-72-75-17
Record Dates: First submitted 2023-01-05; First posted 2023-01-31 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Patellar Dislocation
MeSH Terms: conditions — Patellar Dislocation

STUDY DESIGN:
Intervention Model Description: 1. Standard: Gracillis graft
  2. Intervention: Quadriceps graft
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MPFL reconstruction with gracillis graft (Active Comparator): MPFL reconstructrion with gracillis graft and screw fixation in femur
  Interventions: Procedure: Quadriceps graft
- MPFL reconstruction with quadriceps graft (Experimental): MPFL reconstructrion with quadriceps graft and suture anchor fixation in femur
  Interventions: Procedure: Quadriceps graft

INTERVENTIONS:
Procedure: Quadriceps graft — Using quadriceps graft as new medial patellofemoral ligament graft. Fixated with suture anchor

SUMMARY:
The purpose of this study is to elucidate surgical techniques for reconstructing MPFL in the treatment of chronic patella instability. The two techniques are conventional technique with the gracillis and screw fixation in the femur which is compared with new technique where the QT tendons and anchor fixation in the femur are used.

It would be investigated which technique provides the best stability with the least postoperative pain from the reconstruction and the lowest frequency of patellar reluxation.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 15 and 40 years of age with chronic tendency to lateral patellar dislocation (defined as 2 or more verified dislocation cases)
* The growth zones must be found closed - verified by MRI scan

Exclusion Criteria:

* Patients with known rheumatoid arthritis.
* Patients with arthroscopically detected osteoarthritis (grade 3 cartilage lesion)
* Inability to follow a normal rehabilitation regime.
* Previous ligament surgery in injured knees.

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Kujala (Anterior Knee Pain Scale) | 24 month
  Patient reported outcome score, 0=worst and 100=best

SECONDARY OUTCOMES:
Donor site morbidity score, 0=worst and 100=best | 24 month
  Patient reported outcome score
Knee injury and Osteoarthritis Outcome Score (KOOS) | 24 month
  Patient reported outcome score, 0=worst and 100=best
Lysholm-Tegner (Activity Score) | 24 month
  Patient reported outcome score, 0=worst and 100=best
Numerical Rating Scale (NRS-pain score) | 24 month
  Patient reported outcome score, 0=Best and 10=worst
Knee pain | 24 month
  Palpatory pain in relation to graft fixation in femur on a four-point likert scale (no pain, mild pain, moderate pain, severe pain)
Patella Re-luxation sensation | 24 month
  Question about how often the patella has dislocated after the surgery. (no dislocation, 1-2 dislocation/md, more dislocation).

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Sports Trauma, Palle Juul-Jensens Boulevard 99, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: Undecided